CLINICAL TRIAL: NCT00821028
Title: Treatment of Superficial Femoral Artery Atherosclerotic Disease With Local Delivery of Paclitaxel Using an Irrigating Catheter: a Single-center Pilot Study
Brief Title: Local Paclitaxel Delivery for SFA Disease
Acronym: IRRITAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Atrium-001
Record Dates: First submitted 2009-01-05; First posted 2009-01-12 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Atherosclerosis; Angioplasty; Peripheral Arterial Disease
Keywords: atherosclerosis; angioplasty; peripheral arterial disease
MeSH Terms: conditions — Atherosclerosis; Peripheral Arterial Disease | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel (Experimental): Participants will receive Paclitaxel.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel will be administered intra-arterially through an irrigating catheter to treat a diseased segment of superficial femoral artery. Dosing will be based on ther lesion surface area, and will be calculated using the following formula: dose= 22/7 X diameter (mm) X length (mm) X 3 micrograms/mm^3

SUMMARY:
To see if restenosis rates of superficial femoral artery atherosclerosis with percutaneous techniques can be improved using paclitaxel.

DETAILED DESCRIPTION:
Treatment of superficial femoral artery atherosclerosis with percutaneous techniques is hindered by high restenosis rates. Paclitaxel inhibits restenosis in coronary arteries, and a few studies suggest it may be effective in reducing restenosis rates in peripheral arteries. The investigators hypothesize that delivering paclitaxel through an irrigating catheter will be superior in preventing restenosis.

ELIGIBILITY:
Inclusion Criteria:

* All subjects between 18 and 80 years of age with symptomatic claudication (Rutherford category 1-6) with TASC II type A, B, or C lesions will be invited to participate (23, 24).
* Patients must be on appropriate pharmacologic therapy for PAD including antiplatelet agents and lipid-lowering therapy.

Exclusion Criteria:

* Life expectancy <1year
* Acute limb ischemia
* Anatomy not amenable to percutaneous revascularization
* Inability to provide informed consent
* Renal insufficiency (creatinine clearance <40mL/min calculated using Cockcroft-Gault equation)
* Prisoners
* Pregnant or lactating women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Superficial femoral artery late lumen loss | 12 months

SECONDARY OUTCOMES:
procedural success, amputation, target segment revascularization (TSR), target vessel revascularization (TVR), surgical revascularization, clinical restenosis defined by increase in Rutherford claudication grade of 1 or more | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mazen Abu-Fadel, M.D., Principal Investigator — Univeristy of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States